CLINICAL TRIAL: NCT04931225
Title: LANdiolol MIcrocirculatory Effects During Septic chOc
Brief Title: LANdiolol MIcrocirculatory Effects During Septic chOc (MILANOS)
Acronym: MILANOS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP191047
Record Dates: First submitted 2021-05-14; First posted 2021-06-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Septic Shock
Keywords: Septic shock; Landiolol; Microcirculatory effects; Heart rate; Hemodynamic effects; Microvascular reactivity
MeSH Terms: conditions — Shock, Septic | interventions — landiolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Landiolol injection (Experimental): Intravenous Landiolol injection (from 0.5 to 10 µg/kg/min during 12 hours) up to a 15% decrease in HR on microcirculatory vascular reactivity.
  Interventions: Drug: Landiolol
- Usual tachycardia management (No Intervention): No treatment, usual tachycardia management.

INTERVENTIONS:
Drug: Landiolol — Intravenous Landiolol injection (from 0.5 to 10 µg/kg/min during 12 hours) up to a 15% decrease in HR on microcirculatory vascular reactivity.
  Other Names: Rapibloc
  Arms: Landiolol injection

SUMMARY:
The objectives of this study are to evaluate the effect of continuous intravenous Landiolol injection (from 0.5 to 10 µg/kg/min during 12 hours ) up to a 15% decrease in Heart Rate (HR) on microcirculatory vascular reactivity vs. usual tachycardia management and evaluate the hemodynamic effects of Landiolol vs. usual management in patients with septic shock.

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, open label, evaluation of the efficacy of continuous intravenous Landiolol injection up to a 15% decrease in HR on microcirculatory vascular reactivity vs. usual tachycardia management.

Design:

A monocentric, open-label, randomised, superiority clinical trial

Sample size :

44 patients, 22 in each group

Treatments groups:

Continuous intravenous Landiolol injection ( from 0.5 to 10 µg/kg/min during 12 hours ) up to a 15% decrease in HR on microcirculatory vascular reactivity vs usual tachycardia management

Treatment duration :

24 hours

Assessement:

Landiolol (Rapibloc)'s perfusion will be started at T0 at 0.5 mcg/kg/min and increased by 0.5 mcg/kg/min every 30 minutes in order to achieve a 15% (T1) decrease in HR, within the limit of 10 mcg/kg/min. Then the dosage will be maintained for 2 hours (T2) then the drug will be stopped gradually over 2 hours.

Maximum duration of Landiolol infusion will be 12 hours.

No interim analysis is planned. Analysis will be performed at the end of the study after data review and freezing of database.

ELIGIBILITY:
Inclusion Criteria:

* Sinus tachycardia not compensatory, if the doctor considers that the heart rate acceleration should be treated.
* The study will be carried out in
* reanimated and stabilized septic shock defined as:

  * Septic shock is tachycardic (HR>100/min) patients with sepsis (suspected infection + 2 SOFA points) according to the latest international definition and the need to receive noradrenaline to maintain an average blood pressure above 65 mmHg
  * Patient supported for at least 6 hours, necessary for diagnostic management and hemodynamic optimization according to international standards and for less than 24 hours to limit confounding factors related to prolonged reanimation (sedation) and empowerment of organ failure in general and vascular in particular. Hemodynamic stabilization will be defined as the absence of increased doses of norepinephrine in the previous two hours to limit the risk of hypotension induced by Landiolol infusion.
* Age >18 years
* Patient (or family member) informed consent signature or emergency consent
* Affiliation to a social security system

Exclusion Criteria:

* Asthma
* Patients treated with the following bradycardizing drugs:
* Digitalis
* Bradycardizing calcium channel blockers
* Cordarone
* Other beta-blocker
* Hypersensitivity to Landiolol or to one of its excipients (Mannitol E421, sodium hydroxide)
* Sinus disease
* Cardiogenic shock
* Decompensated heart failure when considered unrelated to arrhythmia
* Pregnant or nursing woman,
* Participation in another interventional research involving the human person or being in the exclusion period following a previous research involving the human person, if applicable
* Ward or curative patient
* Moribund patient
* Estimated life expectancy less than 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of decrease in heart rate (HR) on microcirculatory vascular reactivity | 24 hours
  The objectives of this study are to evaluate the effect of continuous intravenous Landiolol injection (from 0.5 to 10 µg/kg/min during 12 hours ) up to a 15% decrease in HR on microcirculatory vascular reactivity vs. usual tachycardia management in patients with septic shock.

SECONDARY OUTCOMES:
Cardiac flow | 24 hours
  Measure of the cardiac flow to evaluate the hemodynamic effects of Landiolol vs. usual tachycardia management
marbling score | 24 hours
  Measure of the marbling score to evaluate the effects of Landiolol vs. usual tachycardia management
skin recoloration time | 24 hours
  Measure of skin recoloration time to evaluate the effects of Landiolol vs. usual tachycardia management
Arterial lactate clearance | 24 hours
  Measure of sarterial lactate clearance to evaluate the effects of Landiolol vs. usual tachycardia management
Measure of Systemic and endothelial inflammation parameters | 24 hours
  Evaluate the hemodynamic effects of Landiolol vs. usual tachycardia management on Systemic and endothelial inflammation parameters: Plasma cytokines (Procartaplex) VCAM-1 (vascular endothelial cell adhesion molecule), Soluble Endocan (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Hafid AIT-OUFELLA, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Intensive care department, Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided